CLINICAL TRIAL: NCT05634473
Title: A Multicenter, Open-label Study to Evaluate the Sensitivity and Specificity of Inhaled Methacholine in Bronchial Provocation Test
Brief Title: A Study to Evaluate the Sensitivity and Specificity of Inhaled Methacholine in Bronchial Provocation Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TQC3610-CS-01
Record Dates: First submitted 2022-07-18; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with asthma/healthy subjects (Experimental)
  Interventions: Drug: Methacholine Chloride

INTERVENTIONS:
Drug: Methacholine Chloride — Cholinergic agonists

SUMMARY:
A multicenter, open-label study to evaluate the sensitivity and specificity of inhaled methacholine in bronchial provocation test

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following inclusion criteria can be included in this trial:

* 1 Adults 65 years of age ≥ 18 years of age, male or female;
* 2 Normal or abnormal pulmonary function test without clinical significance (FEV1 ≥ 70% predicted);
* 3 Voluntary, signed informed consent, good compliance, can cooperate with the trial observation.

Patients with asthma:

* 4 Clinical diagnosis of asthma patients;
* 5 Patients who can stop using prohibited concomitant drugs (β2 adrenoceptor agonists, anticholinergics, oral bronchodilators, antihistamines, leukotriene receptor antagonists) within the specified period before airway allergic examination;

Healthy subjects:

* 6 Body mass index (BMI) = weight (kg)/height2 (m2), and body mass index is within the range of 18.5 ~ 27.0 (including the critical value).

Exclusion Criteria:

Patients with any of the following criteria will not be included in the trial:

* 1 Patients with a past history of allergy to this type of reagent;
* 2 Patients with a history of heart disease who are difficult to adapt to bronchial provocation test;
* 3 Patients who have undergone thoracic or abdominal surgery within 6 months before the trial;
* 4 Patients who have undergone surgery for intracranial, ophthalmic diseases, ear, nose and throat diseases, and respiratory diseases 6 months before the trial;
* 5 Complicated pneumothorax and other respiratory diseases or tuberculosis and other infectious diseases;
* 6 Patients with diseases that may be affected by the use of cholinergic drugs (epilepsy, bradycardia, coronary artery occlusion, vagal tension, thyroid disease, arrhythmia, peptic ulcer, urinary tract disorders, etc.);
* 7 Patients with a past history of drug dependence or alcohol dependence;
* 8 Previous severe circulatory system diseases, hepatobiliary system diseases, digestive tract diseases, urinary system diseases, kidney diseases, blood diseases, endocrine system diseases, immune system diseases, malignant tumors, etc.;
* 9 Patients who are using cholinase inhibitors (treatment of myasthenia gravis);
* 10 Patients with unexplained urticaria;
* 11 Pregnant and lactating women;
* 12 Subjects with dyspnea, wheezing, wheezing on the day of the trial;
* 13 Patients with myocardial infarction or stroke, combined with hypertension (systolic blood pressure > 200 mmHg, diastolic blood pressure > 100 mmHg);
* 14 Poor cooperation in basic pulmonary function tests, not in line with quality control;
* 15 Use of drugs that will affect airway systolic function and airway inflammation, thereby affecting airway reactivity and can not be discontinued before the test (bronchodilator drugs, glucocorticoids, anti-allergic drugs and triene receptor antagonists and others);
* 16 Current smokers, those who quit for less than one year at the time of screening, and those with a smoking history of more than 10 packs/year;
* 17 Abnormalities in physical examination, laboratory tests, vital signs and test-related tests are clinically significant (based on clinician judgment);
* 18 The investigators think that there are any unsuitable for inclusion;

Patients with asthma:

* 1 Hospitalized for asthma exacerbation within 12 weeks;
* 2 Patients with combined respiratory diseases (such as COPD, etc.) that may affect the efficacy and safety evaluation of the drug;

Healthy subjects:

* 1 Have used any drugs in 2 weeks;
* 2 Patients, immediate family members suffering from allergic diseases (allergic rhinitis, specific rhinitis, allergic conjunctivitis, chronic urticaria, food allergy, etc.);
* 3 Patients with upper respiratory tract infection, acute sinusitis and other infection-related symptoms or have received treatment in 6 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity analysis | On the 1 day of administration
  Sensitivity analysis is percentage of asthmatics subjects with positive final challenge compared with total asthmatics subjects in this study.
Specificity Analysis | On the 1 day of administration
  Specificity is the percentage of healthy subjects with negative results in healthy subjects in this study.
Provocative dose causing a 20% fall (PD20) | On the 1 day of administration
  PD20 is provocative dose causing a 20% fall in forced expiratory volume in 1 second (FEV1) .
Adverse events | Base line to 3 days after dosing
  adverse events occured after administration
heart rate (Vital signs) | Base line to 3 days after dosing
oxyhemoglobin saturation (Vital signs) | Base line to 3 days after dosing
Recovery of forced expiratory volume in 1 second (FEV 1) | Base line to 3 days after dosing
  Recovery of forced expiratory volume in 1 second (FEV 1) after administration to assess safty profile.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Province Hospital of chinese medicine, Guangzhou, Guangdong
  - Liuzhou people's Hospital, Liuchow, Guangxi
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Inner Mongolia Medical Univercity, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Benxi Central Hospital, Benxi, Liaoning
  - Weifang NO.2 People's Hospital, Weifang, Shandong
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou, Zhejiang